CLINICAL TRIAL: NCT05171049
Title: A Multicenter, Randomized, Open-label, Blinded Endpoint Evaluation, Phase 3 Study Comparing the Effect of Abelacimab Relative to Apixaban on Venous Thromboembolism (VTE) Recurrence and Bleeding in Patients With Cancer Associated VTE
Brief Title: A Study Comparing Abelacimab to Apixaban in the Treatment of Cancer-associated VTE
Acronym: ASTER
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anthos Therapeutics, Inc. (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANT-007; 2023-509569-19-00 (Other: EUCT number); CMAA868D12302 (Other: Novartis)
Record Dates: First submitted 2021-11-22; First posted 2021-12-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Venous Thromboembolism; Deep Venous Thrombosis; Pulmonary Embolism
Keywords: Anticoagulants; VTE recurrence rate; PROBE design; LMWH; CAT; Cancer associated VTE; Abelacimab; Apixaban; FXI; Major bleeding events; CRNM bleeding events
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — abelacimab; MAA868; apixaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abelacimab (Experimental): Abelacimab intravenous administration followed by monthly administration of the same dose subcutaneously
  Interventions: Biological: Abelacimab
- Apixaban (Active Comparator): Apixaban administered orally twice a day
  Interventions: Drug: Apixaban

INTERVENTIONS:
Biological: Abelacimab — Abelacimab 150 mg
  Other Names: MAA868
  Arms: Abelacimab
Drug: Apixaban — Apixaban 10 mg followed by 5 mg
  Other Names: Eliquis
  Arms: Apixaban

SUMMARY:
This is a Phase 3,multicenter, randomized, open-label, blinded endpoint evaluation study comparing the effect of abelacimab relative to apixaban on venous thromboembolism (VTE) recurrence and bleeding in patients with cancer associated VTE (ASTER)

DETAILED DESCRIPTION:
Cancer associated thrombosis (CAT) is a severe medical condition which is characterized by high incidence of Venous thromboembolism (VTE) recurrence and high risk for bleeding. The two most common treatments today are low molecular weight heparin (LMWH) and direct anticoagulants (DOACs), in which each has limitations. DOACs are administered orally and are seen as a more convenient alternative though associated with bleeding risk; further, some cancer patients have difficulty swallowing or develop vomiting which leads to unpredictable pharmacodynamic effects with oral therapy. The ANT-007 study will compare treatment with abelacimab monthly administration to apixaban twice daily administration over a 6-month treatment. The study outcomes include VTE recurrence, bleeding event and treatment discontinuation at 6 months

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 years old or other legal maturity age according to the country of residence
* Confirmed diagnosis of cancer (by histology, adequate imaging modality), other than basal-cell or squamous-cell carcinoma of the skin alone with one of the following:

  * Active cancer, defined as either locally active, regionally invasive, or metastatic cancer at the time of randomization and/or
  * Currently receiving or having received anticancer therapy (radiotherapy, chemotherapy, hormonal therapy, any kind of targeted therapy or any other anticancer therapy) in the last 6 months.
* Confirmed symptomatic or incidental proximal lower limb deep vein thrombosis (DVT) (i.e., popliteal, femoral, iliac, and/or inferior vena cava [IVC] thrombosis) and/or a confirmed symptomatic pulmonary embolism (PE), or an incidental PE in a segmental, or larger pulmonary artery.

Patients are eligible within 120 hours from diagnosis of the qualifying VTE

* Anticoagulation therapy with a therapeutic dose of DOAC for at least 6 months is indicated
* Able to provide written informed consent

Exclusion Criteria:

* Thrombectomy, insertion of a caval filter or use of a fibrinolytic agent to treat the current (index) DVT and/or PE
* More than 120 hours of pre-treatment with therapeutic doses of UFH, LMWH, fondaparinux, DOAC, or other anticoagulants
* An indication to continue treatment with therapeutic doses of an anticoagulant other than that VTE treatment prior to randomization (e.g., atrial fibrillation [AF], mechanical heart valve, prior VTE)
* Platelet count <50,000/mm3 at the screening visit
* PE leading to hemodynamic instability (blood pressure [BP] <90 mmHg or shock)
* Acute ischemic or hemorrhagic stroke or intracranial hemorrhage within the 4 weeks preceding screening
* Brain trauma or a cerebral or spinal cord surgery or spinal procedures such as lumbar puncture or epidural/spinal anesthesia within 4 weeks of screening
* Need for aspirin in a dosage of >100 mg/day or any other antiplatelet agent alone or in combination with aspirin
* Primary brain cancer or untreated intracranial metastases at baseline
* Acute myeloid or lymphoid leukemia
* Bleeding requiring medical attention at the time of randomization or in the preceding 4 weeks
* Planned brain, spinal cord, cardiac, vascular, major thoracic and/or major abdominal surgery in the 4 weeks following randomization
* Eastern Cooperative Oncology Group (ECOG) performance status of 3 or 4 at screening
* Life expectancy <3 months at randomization
* Calculated creatinine clearance (CrCl) <30 mL/min (Cockcroft-Gault equation) at the screening visit
* Hemoglobin <8 g/dL at the screening visit
* Acute hepatitis, chronic active hepatitis, liver cirrhosis; or an alanine aminotransferase (ALT) ≥3 x and/or bilirubin ≥2 x upper limit of normal (ULN) at the screening visit in absence of clinical explanation
* Uncontrolled hypertension (systolic BP>180 mm Hg or diastolic BP >100 mm Hg despite antihypertensive treatment)
* Women of child-bearing potential (WOCBP) who are unwilling or unable to use highly effective contraceptive measures during the study from screening up to 3 days after last treatment of apixaban or 100 days after administration of abelacimab (See Section 5.3.6. for highly effective contraceptive measures)
* Sexually active males with sexual partners of childbearing potential must agree to use a condom or other reliable contraceptive measure up to 3 days after last treatment of apixaban or 100 days after administration of abelacimab
* Pregnant or breast-feeding women
* Patients known to be receiving strong dual inducers or inhibitors of both CYP3A4 and P gp
* History of hypersensitivity to any of the study drugs (including apixaban) or excipients, to drugs of similar chemical classes, or any contraindication listed in the label for apixaban
* Subjects with any condition that in the Investigator's judgement would place the subject at increased risk of harm if he/she participated in the study
* Use of other investigational (not registered) drugs within 5 half-lives prior to enrollment or until the expected pharmacodynamic(s) (PD) effect has returned to baseline, whichever is longer. Participation in academic non-interventional studies or interventional studies, comprising testing different strategies or different combinations of registered drugs is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to first event of centrally adjudicated VTE recurrence | Up to 6 months
  Time to first event of centrally adjudicated venous thromboembolism (VTE) recurrence

SECONDARY OUTCOMES:
Time to first event of ISTH-adjudicated major or clinically relevant non-major (CRNM) bleeding events | Up to 6 months
  Time to first adjudicated major or clinically relevant non-major (CRNM) bleeding event
Time to first event of VTE recurrence, ISTH adjudicated major or ISTH-adjudicated clinically relevant non-major (CRNM) bleeding events | Up to 6 months
  Time to first adjudicated venous thromboembolism (VTE) or bleeding event
Time to event of permanent treatment discontinuation not due to death | Up to 6 months
  Time to permanent discontinuation not due to death
Time to first event of ISTH-adjudicated clinically relevant non-major (CRNM) bleeding events | Up to 6 months
  Time to first adjudicated clinically relevant non-major (CRNM) bleeding event
Time to first event of ISTH-adjudicated major bleeding events | Up to 6 months
  Time to first adjudicated major bleeding event
Time to first event of GI ISTH-adjudicated major and CRNM bleeding events | Up to 6 months
  Time to first adjudicated gastrointestinal (GI) major and clinically relevant non-major (CRNM) bleeding event
All-cause death, vascular death, serious adverse events, adverse events leading to drug discontinuation, other adverse events, abnormal lab tests, etc. presented as rate per 100 patient-years | Up to 6 months
For patients treated with abelacimab: percent with injection site reactions/severity, hypersensitivity reactions/severity, anti-drug antibody formation, neutralizing antibody | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (206):
- United States (23):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - Washington DC VAMC, Washington D.C., District of Columbia
  - University of Miami Health, Miami, Florida
  - NorthShore University Health System, Evanston, Illinois
  - University of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center-Middletown, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center-Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center-West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lipson Cancer Institute, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania - Penn Blood Disorders Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Mays Cancer Center, San Antonio, Texas
  - Gundersen Health System, La Crosse, Wisconsin
  - Blood Center of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - Blacktown Hospital, Blacktown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre Clayton, Clayton, Victoria
  - Northern Health, Epping, Victoria
  - Perth Blood Institute, Perth
  - The Alfred Hospital, Prahran
- Austria (3):
  - LKH - Universitätsklinikum Graz, Graz
  - LK Wiener Neustadt, Neustadt
  - Medical University of Vienna, Vienna
- Canada (11):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Hamilton Health Sciences, Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Niagara Health System, Saint Catharines, Ontario
  - Sault Area Hospital, Sault Ste. Marie, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Queen Elizabeth II Health Sciences Centre, Nova Scotia
  - McGill University Health Centre, Québec
- China (13):
  - Beijing Shijitan Hosp., Beijing
  - Peking University Third Hospital, Beijing
  - Jilin Province Tumor Hospital, Ch’ang-ch’un
  - Southern Medical University - Zhujiang Hospital, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - Huizhou Municipal Central Hospital, Huizhou
  - Nanjing First Hospital, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital Tongji Medical College Huazhong University of Science &Technology, Wuhan
  - Tongji Hospital, Tongji Medical College, Wuhan
  - 1st Affiliate Hospital of Xi'an Jiao, Xi'an
- Czechia (5):
  - Masarykuv onkologicky ustav, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - Nemocnice Na Pleši s.r.o., Nová Ves pod Pleší
  - Onkologická klinika VFN a 1. LF UK, Prague
  - Thomayerova nemocnice, Prague
- France (21):
  - CHU Amiens - Hopital Nord, Amiens
  - CHU Angers - Hôpital Hôtel Dieu, Angers
  - CHU de Brest - Hôpital de la Cavale Blanche, Brest
  - CHU Clermont Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Louis Mourier, Colombes
  - CHU Dijon - Hôpital Bocage Central, Dijon
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble
  - CH Le Puy en Velay, Le Puy-en-Velay
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Hopital Timone Adultes, Marseille
  - Centre hospitalier des pays de Morlaix, Morlaix
  - Hôpital Européen Georges Pompidou, Paris
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hospices Civils de Lyon (HCL) - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - CHU de Rouen - Hôpital de Bois Guillaume, Rouen
  - CHU de Saint-Etienne - Hopital Nord, Saint-Etienne
  - CHU Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - Nouvel Hôpital Civil de Strasbourg, Strasbourg
  - Centre Hospitalier Intercommunal de Toulon, Toulon
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
  - CHU de Nancy - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (8):
  - Staedtisches Klinikum Dresden Standort Dresden-Friedrichstadt, Dresden
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Praxis für Gefäßmedizin, Görlitz
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinik der Christian-Albrechts-Universität, Kiel
  - Universitätsklinik Leipzig, Leipzig
  - Universitaetsklinikum Magdeburg A.oe.R, Magdeburg
  - Klinikum der Universitaet Muenchen, München
- Hungary (3):
  - Debreceni Egyetem, Debrecen
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger
  - Bacs-Kiskun County Hospital, Kecskemét
- Ireland (5):
  - Bon Secour Hospital, Cork
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Msdyrt Midericordiae University Hospital, Dublin
  - University Hospital, Limerick, Limerick
- Italy (24):
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Arcispedale S. Maria Nuova Azienda Ospedaliera di Reggio Emilia, Bologna
  - Presidio Ospedaliero di Castelfranco Veneto, Castelfranco Veneto
  - SS. ma Annunziata, Chieti
  - Ospedale Civile Dell Annunziata, Cosenza
  - Ospedale Degli Infermi, Faenza
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Azienda Socio Sanitaria Territoriale Santi Paolo e Carlo, Milan
  - A.O.U. Policlinico di Modena, Modena
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Azienda Ospedale - Università Padova, Padua
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Universit degli Studi di Perugia - Azienda Ospedaliera di Perugia, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Arcispedale S. Maria Nuova Azienda Ospedaliera di Reggio Emilia, Reggio Emilia
  - Fondazione Policlinico Universitario A. Gemelli IRCCS., Roma
  - Istituto Clinico Humanitas, Rozzano
  - Ospedale Santa Maria di Cà Foncello, Treviso
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia, Udine
  - Università dell'Insubria, Varese
  - Ospedale SS. Giovanni e Paolo, Venezia
  - Ospedalemichele e Pietro ferrer, Verduno
  - Ospedale San Bortolo di Vicenza, Vicenza
- Japan (16):
  - National Cancer Center Hospital, Tsukiji, Tokyo
  - Chibaken Saiseikai Narashino Hospital, Chiba
  - Kyushu University Hospital, Fukuoka
  - Tokai University Hospital, Isehara
  - Yokohama Minami Kyosai Hospital, Kanagawa
  - Kobe University Hospital, Kobe
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Mie University Hospital, Mie
  - Tokyo Saiseikai Central Hospital, Minatoku
  - Tohoku University Graduate School of Medicine, Miyagi
  - Okayama Medical Center, Okayama
  - Osaka International Cancer Institute, Osaka
  - International University of Health and Welfare MITA Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Kyorin University Hospital, Tokyo
- Latvia (3):
  - Daugavpils Regional Hospital, Daugavpils
  - Liepaja Regional Hospital, Liepāja
  - Pauls Stradins Clinical University Hospital, Riga
- Netherlands (12):
  - Meander Medisch Centrum, Amersfoort
  - Onze Lieve Vrouwe Gasthuis, Locatie Oost, Amsterdam
  - Rode Kruis Ziekenhuis, Beverwijk
  - Albert Schweitzer Ziekenhuis, Dordwijk, Dordrecht
  - Universitair Medisch Centrum Groningen, Groningen
  - Tergooiziekenhuizen, Hilversum, Hilversum
  - Amsterdam University Medical Center, Holland
  - Spaarne Gasthuis (Kennemer Gasthuis) - Haarlem-Zuid, Hoofddorp
  - Leids Universitair Medisch Centrum, Leiden
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Ikazia Ziekenhuis, Rotterdam
  - Haga Ziekenhuis, The Hague
- Norway (2):
  - Østfold Hospital Kalnes, Fredrikstad
  - Akershus Univeristy Hospital, Lørenskog
- South Korea (11):
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Yongin Severance Hospital, Yonsei University Health System, Yongin-si, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Anyang
  - SoonChunHyang University Hospital Bucheon, Bucheon-si
  - Daegu Catholic University Medical Center, Daegu
  - Jeonbuk National University Hospital, Jeonju
  - Dong-A University Hospital, Seogu
  - Soonchunhyang University Seoul Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Yangcheon
  - Soonchunhyang University Seoul Hospital, Yongsan
- Spain (19):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Del Vinalopo, Elche
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Ciudad de Jaen, Jaén
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - MD Anderson Cancer Centre, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Complejo Hospitalario Universitario de Orense, Ourense
  - Clinica Universidad de Navarra, Pamplona
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario Marques de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
- Länssjukhuset Sundsvall-Härnösand, Sundsvall, Sweden
- Switzerland (3):
  - Hopital Universitaire Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - University of Zürich, Zurich
- Taiwan (8):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Tri-Service General Hospital, Taipei
- United Kingdom (7):
  - University Hospital of Wales, Cardiff, England
  - University Hospitals of North Midlands, Stafford, England
  - University Hospitals of North Midlands, Stoke-on-Trent, England
  - Castle Hill Hospital, Department of Oncology & Haematology, Cottingham, ENG
  - Barts Health NHS Trust, London, ENG
  - The Newcastle Upon Tyne Hospitals, Newcastle upon Tyne, ENG
  - Queen Elizabeth University Hospital Campus, Glasgow, SCO

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com